CLINICAL TRIAL: NCT07078448
Title: The Sex-Specific Impact of a Single Foam Rolling Session on Peripheral Muscle Oxygenation in Recreational Adults With Hamstring Tightness
Brief Title: The Sex-Specific Impact of a Single Foam Rolling Session on Peripheral Muscle Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pelin Pişirici (Other)
Responsible Party: Sponsor-Investigator, Pelin Pişirici, Assistant Professor, PT, PhD, Bahçeşehir University
Organization: Bahçeşehir University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GP-FR-25G
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hamstring Muscles; Hamstring Shortness; Hamstring Tightness
Keywords: Moxy; Myofascial Release; hamstring shortness; Near-Infrared Spectroscopy; range of motion

STUDY DESIGN:
Intervention Model Description: Participants who met the inclusion criteria were divided into two groups according to sex (female and male). Each group received the same foam roller intervention. Hamstring muscle oxygenation and joint range of motion were measured before the intervention, immediately after, and ten minutes post-intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- female (Experimental): foam roller intervention
  Interventions: Other: Foam Roller
- male (Experimental): foam roller intervention as the females received
  Interventions: Other: Foam Roller

INTERVENTIONS:
Other: Foam Roller — FR will be applied to each hamstring muscle for 3 minutes per leg, totaling 6 minutes. The pressure was self-regulated by participants, who are instructed to apply as much body weight as tolerable. The rolling frequency is maintained at approximately 0.5 Hz, corresponding to one complete rolling cycle every 2 seconds. Before the intervention, participants will receive verbal and visual instructions to ensure correct execution.

SUMMARY:
The hamstring muscle, as a biarticular muscle, plays a crucial role in both hip extension and knee flexion and is part of the Superficial Back Line, which supports upright posture and prevents excessive flexion. Its continuous postural function requires endurance-oriented muscle fibers and sustained low-level muscle tone. Tightness in the hamstrings is commonly linked to postural imbalances and structural factors, contributing to gait alterations, low back pain, tendinopathy, and other musculoskeletal disorders. Improving hamstring flexibility is important for performance and injury prevention, with myofascial release-particularly self-myofascial release using foam rollers-being an effective method. Foam rolling reduces muscle tension, enhances tissue hydration, and may alleviate fascial adhesions. However, sex differences exist in connective tissue properties, potentially influencing outcomes. Limited research has explored foam rolling's impact on peripheral muscle oxygenation. This study aims to investigate the effect of foam rolling on hamstring muscle oxygen saturation in recreational individuals with tightness, with a hypothesis that females may show greater increases.

DETAILED DESCRIPTION:
The hamstring muscle is a biarticular muscle that simultaneously contributes to both hip extension and knee flexion movements. From the perspective of myofascial continuity, the hamstring is part of the Superficial Back Line, whose general postural function is to support the body in a fully upright position and to prevent the tendency toward flexion. This continuous postural role throughout the day necessitates a higher proportion of slow-twitch, endurance-oriented muscle fibers within the muscular segments of this myofascial chain. The hamstrings, as components of this line, maintain a low-level but sustained tone during the day to support posture.

Tightness in the hamstring muscles frequently arises due to issues in structural connectivity such as segmental shortening or tension along the Superficial Back Line, prolonged postural loading, imbalances with the Superficial Front Line, or alterations in pelvic tilt. It has been demonstrated that hamstring tightness can lead to alterations in gait patterns, low back pain, patellar tendinopathy, plantar fasciitis, and hamstring injuries.

Hamstring flexibility is a fundamental factor for individuals to enhance their sports performance and maintain a healthy lifestyle. Achieving adequate range of motion or flexibility not only supports the optimal functioning of the musculoskeletal system but also contributes to the prevention of injuries and muscular imbalances. One of the methods employed to improve hamstring flexibility is myofascial release. According to a meta-analysis examining the immediate effects of myofascial release applied along the Superficial Back Line in adults, the majority of studies have reported improvements in joint range of motion (ROM) and muscle flexibility.

One technique known as self-myofascial release is the use of a foam roller. A foam roller is a rigid cylindrical tool made of foam, available in various densities and sizes. The pressure applied with a foam roller stimulates the Golgi tendon organ, thereby reducing muscle tension. Another possible effect is the enhancement of tissue hydration; during application, the soft tissues are compressed like a sponge, allowing fluids to permeate the tissues, facilitating movement between fascial layers, and increasing blood flow and tissue temperature. Additionally, it is hypothesized that foam rolling helps release fascial adhesions and reduces scar tissue formation.

The physiological properties of connective tissues differ between males and females. Women are generally considered to be more flexible compared to men and structurally demonstrate greater tissue compliance, exhibiting a higher capacity to stretch or adapt to deformation. Therefore, the effects observed following foam roller application may vary between sexes. One study sought to investigate the sex-specific effects of acute self-myofascial release on joint range of motion and muscle stiffness. Following a foam roller intervention consisting of two sets of 30 seconds, no significant difference was observed in soft tissue stiffness or joint range of motion among female participants; however, significant improvements were noted in the male group regarding plantar flexion, dorsiflexion, and plantar flexion range of motion. Analysis of covariance comparing sex differences revealed significant differences between groups in the medial region of the Achilles tendon and gastrocnemius muscle. These findings suggest that short-duration self-myofascial release sessions may be sufficiently effective in increasing ankle joint range of motion in males; however, further research is needed to generalize these results to females. Due to inconclusive findings regarding soft tissue stiffness across sexes, larger sample sizes are recommended to explore this topic further.

It is known that a single session of foam rolling can increase flexibility and joint range of motion; however, studies investigating the effect of foam rolling on peripheral muscle oxygenation remain limited. One study examined the effects of four different interventions-dynamic stretching combined with foam rolling, static stretching combined with foam rolling, static stretching alone, and eccentric exercise alone-on fascicle length, muscle-tendon unit stiffness, muscle oxygen saturation (SmO₂), and muscle performance. The results indicated a tendency for SmO₂ levels to decrease following eccentric exercise, while immediate increases were observed in the other three interventions. However, this research was not sex-specific and did not isolate the effect of foam rolling on the SmO₂ of the hamstring muscle.

The aim of the present study is to investigate the effect of foam rolling on muscle oxygen saturation of the hamstring muscle in recreational individuals with hamstring tightness. Our hypothesis is that muscle oxygenation will increase to a greater extent in females.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged between 18 and 35 years
* Both male and female participants
* Absence of any known health conditions
* Hamstring tightness defined as ≥20° of knee flexion angle in Active Knee Extension test

Exclusion Criteria:

* Any neuromuscular or orthopedic disorders affecting the lower extremities
* Circulatory or vascular problems
* Respiratory or cardiovascular diseases
* Renal failure
* Presence of pain during measurements or exercise protocols
* Excessive skin sensitivity or active skin infection
* History of intense physical activity within the last 48 hours

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — No, gender identity did not differ from biological sex in any participant; therefore, eligibility was based on biological sex.
Enrollment: 36 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Muscle Oxygenation Assessment | baseline, immediately after the intervention, ten minutes after the baseline
  Muscle oxygenation will be assessed using the MOXY Monitor, a portable, wireless, near-infrared spectroscopy (NIRS)-based device. The monitor will be placed on the belly of the right biceps femoris muscle and secured with an opaque elastic band to prevent ambient light interference.
  Measurements will be taken five minutes before and five minutes after the intervention session. During each measurement, the device will record data for 60 seconds, and the average SmO₂ (muscle oxygen saturation) value over this period will be used for analysis.

SECONDARY OUTCOMES:
Active Knee Extension (AKE) Test | baseline, immediately after the intervention, ten minutes after the baseline
  The AKE test will be used as a secondary outcome measure to assess hamstring flexibility. Participants will lie supine with the non-tested leg extended. The tested leg will be positioned in 90° of hip flexion using a wooden box to stabilize the pelvis and thigh.
  Participants will actively extend the knee until a visible myoclonus occurs. They will then slowly lower the leg until the movement stops. At that point, the knee flexion angle will be measured using a goniometer. The average of three trials will be recorded for each leg.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Koçak, MD, Principal Investigator — Medipol University; Pelin Pişirici, PT, PhD, Study Chair — Bahcesehir University, Faculty of Health Sciences
Locations (1):
- Bahçeşehir University, Istanbul, Beşiktaş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No